## **Informed Consent Form**

Official Title: A Story-Based Digital Game to Reduce Anxiety and Improve Treatment

Compliance in Hemodialysis Patients: A Randomized Controlled Trial

NCT Number: To be assigned

**Ethics Committee Approval Number:** E.888577

**Study Period:** March 2025 – April 2025

## INFORMED CONSENT FORM Participant Information and Consent Form

Dear Participant,

We are conducting a study to evaluate the use and impact of a story-based digital game for hemodialysis patients. The study is titled: "A Story-Based Digital Game to Reduce Anxiety and Improve Treatment Compliance in Hemodialysis Patients: A Randomized Controlled Trial."

You are invited to participate in this study. Your participation is entirely voluntary. Before you decide whether to participate, we would like to inform you about the study's purpose, process, and your rights as a participant. The aim of this study is to evaluate the effects of a story-based digital game developed for hemodialysis patients on reducing anxiety levels, improving treatment adherence, and increasing dietary knowledge.

This study will be conducted between March and April 2025 with patients who regularly attend the Hemodialysis Unit at Suleyman Demirel University Research and Training Hospital. It is a randomized controlled study comparing two groups. Participants will be randomly assigned to either the control group, which receives standard care, or the intervention group, which will use the story-based digital game in addition to standard care. Those in the intervention group will play the digital game during one dialysis session for approximately 10–15 minutes. Data will be collected from all participants before and after the intervention using the following scales: State Anxiety Scale, Hemodialysis Patients' Diet Knowledge Scale, and End-Stage Renal Disease Adherence Scale.

Your participation is entirely voluntary. You may withdraw from the study at any time without any consequences or impact on your medical treatment. You will not receive any compensation for participating, and there are no financial costs involved. Your identity will remain confidential, and your data will only be used for scientific purposes anonymously.

| If you have any questions about the study, please contact: |
|---|
| I have read and understood the information provided above. All my questions were answered |
| clearly. I voluntarily agree to participate in this study. |

| Participant Name: | | _ |
|-------------------|---------|---|
| Signature: | Date: _ | |